CLINICAL TRIAL: NCT06212206
Title: Feasibility and Safety of PillBot™ - Remotely Controlled Capsule Endoscopy: A Feasibility Study
Brief Title: PillBot™ - Remotely Controlled Capsule Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Endiatx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Endiatx
Record Dates: First submitted 2023-12-26; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Gastric Disease
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PillBot (Experimental): Patient will swallow the PillBot and be assessed with EGD after two hours of the examination
  Interventions: Device: PillBot

INTERVENTIONS:
Device: PillBot — The PillBot System uses active, motorized propulsion technology to facilitate the navigation and positioning of the capsule within the stomach anatomy for imaging of the gastric mucosa by an operator.

SUMMARY:
The PillBot System is an endoscopic capsule imaging system intended for visualization of the stomach. In contrast to currently used passive capsule endoscopy systems, and FDA cleared active magnetic system, the PillBot System uses active, motorized propulsion technology to facilitate the navigation and positioning of the capsule within the stomach anatomy for imaging of the gastric mucosa by an operator

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ability to provide written, informed consent to undergo both capsule endoscopy (un-sedated) and conventional OGD
* Willing and able to complete study follow-up requirements
* Patient has appropriate indications for upper endoscopy including symptoms of, but not limited to upper abdominal pain, acid reflux, heartburn, iron deficiency anemia, weight loss, bloating, belching, nausea, vomiting and atypical chest pain

Exclusion Criteria:

All patients who meet any of the following criteria should not be enrolled into the study:

* Coagulopathy with INR > 1.5, thrombocytopenia with platelet counts < 50,000
* Active bleeding
* Need for therapeutic procedures during endoscopy
* Lactation
* Dysphagia, or other swallowing disorders
* Known esophageal diverticulum or stricture
* Swallowing disorder
* Known luminal, gastrointestinal strictures
* Patient with Crohn's disease or other potential obstructive conditions, unless there is a recent Computed tomography enterography (CTE) or Magnetic resonance enterography (MRE), MRE or patency capsule performed to exclude an obstructive lesion that may retain the capsule
* History of esophageal, gastric surgery or intestinal surgery
* Esophageal or GI motility disorder
* Known or suspected gastrointestinal obstruction, significant intestinal strictures, or fistulas based on the clinical picture or pre-procedure testing and profile.
* Current participation in another investigational drug or device treatment study
* Pregnant or wishes to become pregnant during the study follow-up period
* Patient with implanted medical device that would be potentially affected radiofrequency emissions (e.g., pacemakers, implanted cardiac defibrillators)
* Severe psychiatric, neurological, cardio-vascular, or renal disorders
* History of allergy or intolerance to materials used to make the PillBot

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | Up to two weeks
  Adverse events rate during and following device use.
Primary Effectiveness Endpoint | Through study completion, an average of two weeks
  Identification of the gastric anatomy landmarks (cardia, fundus, body, angulus, antrum, and pylorus) with PillBot compared to conventional endoscopy.

SECONDARY OUTCOMES:
Secondary Study Endpoints | Through study completion, an average of two weeks
  1. Complete gastric examination using PillBot and its passage into the duodenum.
  Complete gastric examination is defined as the ability to identify and distinguish lesion type (i.e., polyps, ulcers, submucosal humps, etc.), lesion size (e.g., <5mm and > 5mm) and location when using the PillBot compared with conventional endoscopy.
Secondary Study Endpoints | Through study completion, an average of two weeks
  2. Accuracy of gastric lesions detection by the RCE compared to the upper endoscopy based on independent reviewer's assessment.